CLINICAL TRIAL: NCT02398331
Title: Impact of an Information and Education Program on Sexuality and Social Integration in Women With a Spinal Cord Injury
Brief Title: Sexual Health of Spinal Cord Injured Females
Acronym: SexSIFem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P130912
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2017-11

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; Sexual function; Sexual response; Sexuality; Women
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm (Experimental): Standardised information and education on sexuality in women with spinal cord injury
  Interventions: Other: Standardised information and education on sexuality in women with spinal cord injury
- Control arm (No Intervention): Usual care (no structured information or education on sexuality)

INTERVENTIONS:
Other: Standardised information and education on sexuality in women with spinal cord injury — Program of information and education on the physiology of sexual response in women with spinal cord injury 6 months after their first return to home:
  * Educational footage
  * Clinical neurological examination with educational aim
  * Structured consultation providing information on the physiology of sexual response in women with spinal cord injury
  Arms: arm

SUMMARY:
The purpose of this study is to assess the impact on sexuality in women with a spinal cord injury, twelve months after their first return to home, of a program including structured information and education on sexuality, delivered 6 months after their first return to home.

DETAILED DESCRIPTION:
Multicentre, prospective study, aiming to assess the effect on sexuality of an information and education program in women with spinal cord injury.

Included patients will be women hospitalized for initial rehabilitation, and will be included two weeks before their first return to home.

Socio-demographic data, diagnosis and etiology, secondary conditions, treatment, comorbidities and expectations towards rehabilitation care will be assessed at inclusion.

At M3 Patients will be randomized in either the intervention arm or the control arm.

Patients enrolled in the intervention arm will benefit from a standardised information and education consultation on physiology of sexual response 6 months after their return home.

Patients enrolled in the control arm will undergo the same follow-up but will only have the usual unstructured and unformalized information provided by the clinical team.

At M3, M6, M12 secondary conditions , sexual function index (FSFI), social integration (LHS), treatment and expectations towards rehabilitation care will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury including cauda equina injury of traumatic etiology or not
* Hospitalization for initial post-injury rehabilitation in a study center
* First return at home scheduled within the 14 days following inclusion date
* Understanding of the French language allowing to answer questionnaires
* Affiliation to health insurance
* Written informed consent

Exclusion Criteria:

* Full recovery of sensory-motor functions (AISE)
* Associated brain injury
* Psychiatric disease previously diagnosed, excepted treated and remitting mood disorders
* Patients with tutorship / guardianship
* Spinal cord injury of malignant origin
* Spinal cord injury associated with multiple sclerosis
* Anticipated loss-to-follow-up (patient moving outside of the usual hospital catchment area)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) 12 months after returning home | 12 months

SECONDARY OUTCOMES:
Hospital anxiety and depression scale (HAD) | 12 months
London Handicap Scale (LHS) | 12 months
Expectations of women in terms of care | 12 months
Stability or change of sexual partner | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François Giuliano, MD, PhD, Principal Investigator — Physical and Rehabilitation Medicine Department, Raymond Poincaré Hospital, 92380 Garches, France
Locations (1):
- Physical and Rehabilitation Medicine Department, Raymond Poincaré Hospital, Garches, Hauts-de-Seine, France